CLINICAL TRIAL: NCT06261463
Title: Leveraging Implementation Science and Design Methods to Sustain Community-based Mental Health Services for Refugees
Brief Title: Hybrid Type 1 Randomized Pilot Trial of a Peer-led Family and Social Strengthening Group Intervention for Refugee Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mary Bunn, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-0326; K01MH128524-01A1 (NIH)
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Depression; Anxiety; PTSD; Family Dynamics; Social Functioning; Family Support; Family Relations
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Social Adjustment | interventions — Coffee; Palliative Care

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a randomized controlled trial with refugee families from Arabic-speaking refugee families from the Middle East (n=74). Half of the participants will be randomized to receive CAFES2 and half will be randomized to the enhanced control condition where they will receive ongoing access to services through partner organizations and healthy lifestyle materials.
Who Masked: Outcomes Assessor
Masking Description: The Research Assistants (RAs) who will collect both qualitative and quantitative data will be blind to the condition in which study participants are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAFES2 family and social strengthening intervention (Experimental): Families randomized into CAFES2 receive a home visit and participate in six multiple family group sessions in addition to any outside services or programs they are participating in.
  Interventions: Behavioral: CAFES2
- Enhanced Control (No Intervention): Families randomized to the enhanced control arm will not receive the CAFES2 intervention Instead, they will continue with their usual care, and also receive healthy lifestyle materials.

INTERVENTIONS:
Behavioral: CAFES2 — The adapted CAFES2 model includes an initial home visit and six multiple family group sessions delivered by peer providers. Families include at least one caregiver and one youth 12 years or older. Key model components include: 1) interfamilial discussion of stressors affecting families and family relationships, 2) psychoeducation on the effects of war and forced displacement on individuals, families and social relationships; 3) emotion regulation and self management strategies; 4) identification and activation of family and social strengths, 5) discussion of family identity and hopes for the future in resettlement and 5) discussion of social and community resources to support health and wellbeing. Each group session incorporates didactic components, family and small group discussion, skill building and separate breakout groups for adolescents and adults.
  Other Names: Coffee and Family Education and Support, Version 2
  Arms: CAFES2 family and social strengthening intervention

SUMMARY:
The proposed study draws on prior research to evaluate the feasibility, acceptability and explore preliminary effectiveness of Coffee and Family Education and Support, Version (CAFES2) using a pilot randomized type 1 hybrid effectiveness-implementation design. CAFES2 is a peer-led family and social strengthening multiple family group intervention that is designed to respond to multi-level needs of refugee families. Results of the trial will contribute to the emerging evidence base on family-based mental health interventions for refugee and newcomer communities. The trial will also generate new insights regarding implementation strategies needed to promote successful delivery of services by peer providers and the unique role of human-centered design practices for adaptation of mental health and psychosocial interventions.

DETAILED DESCRIPTION:
In partnership with refugee service organizations in Chicago, the investigator explored the problems, strengths, and help-seeking preferences of refugee families. Qualitative findings indicated ongoing problems coping with stress, trauma and loss, strain and tension in family relationships and limited social support networks. Participants identified a need for family-focused, group-based services led by individuals with similar life experiences. Based on these findings, the investigators identified an evidence-based multiple-family group model, Coffee and Family Education and Support (CAFES) as a foundational model that could be adapted to meet the needs of refugee families. Drawing on this formative work and strong community partnerships, further research is needed to adapt CAFES to a new population, to reflect multi-level needs of families and for use by refugee peer facilitators in community-based organizations. Research is also needed to assess feasibility, acceptability and fidelity of model implementation, attentive to barriers and facilitators specific to peer-led mental health services and community settings.

The investigators will use a hybrid type 1 randomized pilot trial design to achieve the following specific research aims:

Aim 1: To adapt the multiple family CAFES model for delivery by peers in community organizations using an implementation science adaptation framework and participatory human-centered design methods to develop an intervention that addresses the complex needs of refugee families.

Aim 2: To pilot the adapted CAFES2 model with refugee families from Arabic-speaking countries in the Middle East to examine feasibility, acceptability and provider fidelity when implemented by refugee peers in two community-based organizations in Chicago. (n=74, 37 intervention, 37 control) Aim 3: To explore the impact of the adapted CAFES2 model compared to enhanced control on outcomes of adult and child mental health and family and community support and explore variables expected to mediate the intervention's impact.

ELIGIBILITY:
To participate in the study, the families must meet the following criteria:

1. Country of origin: Iraq, Syria, Lebanon, Jordan, Palestine or Yemen
2. refugee family living in Chicago < three years
3. Contains at least one adult caregiver (18-55) and at least one of their children (age 12 and older) living in one household
4. One family member with > 3 on the GHQ-12
5. able to give written informed consent.

Exclusion criteria for refugee families:

1. Not from one of the following Arabic-speaking countries in the Middle East: Iraq, Syria, Jordan, Lebanon, Palestine, Yemen
2. men and women who do not have least one child aged 12 years and older living in one household
3. arrived in the U.S as a refugee greater than 3 years ago
4. persons with developmental disabilities which would preclude their participation in the adapted CAFES intervention
5. persons with severe mental health (e.g., suicidality psychotic disorder), active substance use or current in family crisis (e.g., domestic violence, divorce proceedings).

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in feasibility of the intervention via the Feasibility of Intervention Measure | immediate post-intervention
  This 4-item measure assesses the degree to which a given intervention is viewed as feasible for a given population and setting. Higher scores are associated with greater degrees of perceived feasibility.
Changes in acceptability of the intervention via the Acceptability of Intervention Mesure | immediate post-intervention.
  4-item measure assess the degree to which the intervention is viewed as agreeable or satisfactory, with higher scores indicating greater acceptability
Changes in PTSD symptoms via the PTSD Checklist (adult, exploratory) | baseline, immediate post-intervention and 6-week follow up
  PTSD Checklist utilizes a 5-point likert scale (0-4) to assess post traumatic stress symptoms. Higher scores indicate increasing levels of PTSD.
Changes in adult depression and anxiety via the Hopkins Symptom Checklist (HSCL, adult, exploratory) | baseline, immediate post-intervention and 6-week follow up
  HSCL measures symptoms of anxiety and depression in adults using a 4-point likert scale (1-4) with high scores indicating higher levels of anxiety and depression symptoms.
Changes in youth depression and anxiety via the Arab Mental Health Scale (youth, exploratory) | baseline, immediate post-intervention and 6-week follow up
  This scale measures symptoms of anxiety and depression in youth using a 3-point likert scale (0-3). Total scores are associated with mild, moderate or severe anxiety or depression.
Changes in PTSD in children and youth via the Child Revised Impacted of Events Scale (CRIES, youth, exploratory) | baseline, immediate post-intervention and 6-week follow up
  CRIES is a measures to assess PTSD symptoms in children and youth. Higher total scores indicate higher PTSD symptoms.
Changes in post-migration stress in youth and adults via the Refugee Post-Migration Stress Scale | baseline, immediate post-intervention and 6-week follow up
  The post-migration stressors scale assess stress in youth and adults. Higher total scores indicate higher levels of stress.

SECONDARY OUTCOMES:
Changes in social support via the Medical Outcomes Study (MOS) Social Support Survey | baseline, immediate post-intervention and 6-week follow up
  This measure assesses diverse forms of social support using a 5-point likert scale. Higher overall scores indicate greater degree of available support.
Changes in social interaction via the Duke Social Support Index, social interaction subscale | baseline, immediate post-intervention and 6-week follow up
  The Duke Social Support Index, Social Interaction Subscale assesses diverse types of daily social interactions. Higher scores indicate greater degrees of social interaction.
Changes in family support via the Multidimensional Scale of Perceived Social Support (MSPSS, Family Support Sub-scale) | baseline, immediate post-intervention and 6-week follow up
  Likert scale (1-7) that assesses degree of family support. Higher scores indicate greater degress of family support.
Quality of the parent-child relationship via the Dimensions of Parenting Scale (sub-scale, warmth and responsiveness of parent-child relationship) | baseline, immediate post-intervention and 6-week follow up
  The Dimensions of Parenting, Warmth and responsiveness sub-scale assess the nature and quality of the parent-child relationship using a 3-point likert scale (1-3). Higher scores indicate greater degree of parent-child warmth and responsiveness.
Degree of family strengths and difficulties via the SCORE-15 (family strengths, family difficulties sub-scales | baseline, immediate post-intervention and 6-week follow up
  A 15-item scale assess family communication, strengths and difficulties with lower scores indicating higher levels of family strengths and higher scores more family difficulties

CONTACTS AND LOCATIONS:
Overall Officials: Mary Bunn, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinios Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No